CLINICAL TRIAL: NCT00513656
Title: A Randomised, Double-blind, Active-controlled, Double-dummy, Parallel Group Study to Determine the Safety and Efficacy of Oxycodone/Naloxone Prolonged Release Tablets in Subjects With Moderate to Severe, Chronic Cancer Pain
Brief Title: A Study Comparing Oxycodone to Oxycodone/Naloxone in Moderate to Severe, Chronic Cancer Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mundipharma Research GmbH & Co KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OXN2001; 2007-001313-42
Record Dates: First submitted 2007-07-27; First posted 2007-08-09 (Estimated); Last update posted 2018-10-23 (Actual); Status verified 2012-08

CONDITIONS: Cancer; Pain; Constipation
Keywords: Efficacy; chronic; cancer; pain; constipation; oxycodone; naloxone; Moderate to severe chronic cancer pain
MeSH Terms: conditions — Neoplasms; Pain; Constipation; Bronchiolitis Obliterans Syndrome | interventions — Oxycodone; Naloxone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxycodone Hydrochloride Tablets (Active Comparator)
  Interventions: Drug: Oxycodone
- Oxycodone Naloxone Tablets (Experimental)
  Interventions: Drug: Oxycodone/Naloxone

INTERVENTIONS:
Drug: Oxycodone
  Arms: Oxycodone Hydrochloride Tablets
Drug: Oxycodone/Naloxone
  Arms: Oxycodone Naloxone Tablets

SUMMARY:
The purpose of this study is to test the oxycodone/naloxone combination compared to oxycodone alone in patient's specific type of "chronic cancer pain".

DETAILED DESCRIPTION:
This is a randomised, double-blind, active-controlled, double-dummy, parallel group study using oxycodone/naloxone and oxycodone to treat moderate to severe, chronic cancer pain. Subjects with documented history of cancer pain that requires around-the-clock opioid therapy will be included. Subjects must have a medical history of constipation that was induced by, or worsened by their opioid therapy.

After subjects have qualified for the study they will be randomised and to enter the double-blind treatment phase of the study.

Subjects will be randomised to receive either oxycodone/naloxone or oxycodone. Subjects will receive the double-blind medication for a period of 4 weeks.

Subjects who complete the double-blind phase or who discontinue due to constipation and still comply with all relevant screening inclusion and exclusion criteria will have the option to enter the 24 week extension phase. Subjects will receive open-label oxycodone/naloxone for up to 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects at least 18 years or older with a diagnosis of cancer.
2. Females less than one year post-menopausal must have a negative urine pregnancy test recorded at the screening visit, be non-lactating, and willing to use adequate and highly effective method of contraception throughout the study. Highly effective methods of birth control are defined as those which result in a low failure rate (i.e. less than 1% per year) when used consistently and correctly such as sterilization, implants, injectables, combined oral contraceptives, some IUDs (hormonal), sexual abstinence or vasectomised partner.
3. Subjects who are receiving WHO step II or Step III analgesic medication who have constipation induced, or worsened by their opioid medication, as shown by

   1. the subject's medical need of regular intake of laxatives to have at least 3 bowel evacuations per week, or having less than 3 bowel evacuations when not taking a laxative, respectively.
   2. the subject's self-assessment that their constipation was induced or worsened by their current pre-study opioid medication.
4. Documented history of moderate to severe, chronic cancer pain that requires around-the-clock opioid therapy (starting dose at the beginning of the double-blind phase of oxycodone PR between 20 - 80 mg/day) and are likely to benefit from WHO step III opioid therapy for the duration of the study. Subjects must be willing to discontinue their current opioid analgesic routine.
5. Subjects are willing to discontinue pre-study laxative medication and take study specific laxative medication.
6. Subjects taking daily fibre supplementation or bulking agents are eligible if they can be maintained on a stable dose and regimen throughout the study, and in the investigators opinion are willing and able to maintain adequate hydration.
7. Subjects willing and able (e.g. mental and physical condition) to participate in all aspects of the study, including use of medication, completion of subjective evaluations, attending scheduled clinic visits, completing telephone contacts, and compliance with protocol requirements as evidenced by providing written, informed consent.
8. Subjects already taking non-opioid analgesics and all other concomitant medications (including those for the treatment of depression) are eligible to take part in the study. However, all concomitant medications that are considered necessary for the subject's welfare should be continued at a stable dose throughout the double-blind phase of the study and under the supervision of the investigator. Regarding cyclic chemotherapy please see exclusion criteria list.

Exclusion Criteria:

1. Subjects that require a dose >80 mg/day oxycodone PR at the start of the double-blind phase.
2. Any history of hypersensitivity to oxycodone, naloxone, bisacodyl, related products, and other ingredients.
3. Subjects with any situation in which opioids are contra-indicated, severe respiratory depression with hypoxia and/or hypercapnia, severe chronic obstructive pulmonary disease, cor pulmonale, severe bronchial asthma, paralytic ileus.
4. Evidence of clinically significant cardiovascular, renal, hepatic or psychiatric disease, as determined by medical history, clinical laboratory tests, ECG results, and physical examination, that would place the subject at risk upon exposure to the study medication or that may confound the analysis and/or interpretation of the study results.
5. Abnormal aspartate aminotransferase (AST; SGOT), alanine aminotransferase (ALT; SGPT), or alkaline phosphatase levels (>3 times the upper limit of normal) or an abnormal total bilirubin and/or creatinine level(s) (greater than 1.5 times the upper limit of normal).
6. Subjects with known or suspected unstable brain metastases or spinal cord compression that may require changes in steroid treatment throughout the duration of the study.
7. Subjects with uncontrolled seizures.
8. Subjects with increased intracranial pressure.
9. In the investigator's opinion, subjects who are receiving hypnotics or other central nervous system (CNS) depressants that may pose a risk of additional CNS depression with opioid study medication.
10. Subjects with myxodema, not adequately treated hypothyroidism or Addisons disease.
11. Active alcohol or drug abuse and/or history of opioid abuse.
12. Subjects receiving opioid substitution therapy for opioid addiction (e.g. methadone or buprenorphine).
13. Subjects with evidence of clinically significant gastrointestinal disease (e.g. paralytic ileus, peritoneal carcinosis), significant structural abnormalities of the gastrointestinal tract (e.g. scarring, obstruction etc) either related or not related to the underlying cancer or disease progression.
14. Subjects who have a confirmed diagnosis of ongoing irritable bowel syndrome.
15. Subjects suffering from diarrhea and/or opioid withdrawal.
16. Surgery completed prior to the start of the Screening Period, or planned surgery during the study that would influence pain or bowel function during the study or preclude completion of the study.
17. Cyclic chemotherapy in the two weeks before the screening visit or planned during the core study that has shown in the past to influence bowel function. If subjects are having their first cycle of chemotherapy during the 2 weeks before the screening visit or during the double-blind phase of the study they should be excluded from the study.
18. Radiotherapy that, in the investigators opinion, would influence bowel function or pain during the double-blind phase of the study.
19. Subjects presently taking, or who have taken, naloxone 30 days prior to the start of the Screening Period.
20. Subjects who participated in a clinical research study involving a new chemical entity or an experimental drug within 30 days of study entry (defined as the start of the Screening Period).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2007-09; Primary Completion 2010-03 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Efficacy variable: Bowel Function Index (BFI) score. Amount of laxative medication use recorded at each assessment visit | 4 weeks and a 6 month open label
Efficacy variable: Brief Pain Inventory Short-Form (BPI-SF) (Cleeland, 1991). Amount of analgesic rescue medication used | 4 weeks and a 6 month open label

SECONDARY OUTCOMES:
Number of bowel movements
Modified Subjective Opiate Withdrawal Scale (SOWS)
EuroQol EQ-5D
EORTC QLQ-C30
PAC-SYM
PAC-SYM(b)

CONTACTS AND LOCATIONS:
Overall Officials: Sam Ahmedzai, Principal Investigator — University of Sheffield
Locations (1):
- Dr S Ahmedzai, Sheffield, United Kingdom

REFERENCES:
- [Derived] Koopmans G, Simpson K, De Andres J, Lux EA, Wagemans M, Van Megen Y. Fixed ratio (2:1) prolonged-release oxycodone/naloxone combination improves bowel function in patients with moderate-to-severe pain and opioid-induced constipation refractory to at least two classes of laxatives. Curr Med Res Opin. 2014 Nov;30(11):2389-96. doi: 10.1185/03007995.2014.971355. Epub 2014 Oct 13. PMID 25265132
- [Derived] Ahmedzai SH, Nauck F, Bar-Sela G, Bosse B, Leyendecker P, Hopp M. A randomized, double-blind, active-controlled, double-dummy, parallel-group study to determine the safety and efficacy of oxycodone/naloxone prolonged-release tablets in patients with moderate/severe, chronic cancer pain. Palliat Med. 2012 Jan;26(1):50-60. doi: 10.1177/0269216311418869. Epub 2011 Sep 21. PMID 21937568
- See also: Results available on website — https://www.clinicaltrialsregister.eu/ctr-search/search?query=OXN2001